CLINICAL TRIAL: NCT04009109
Title: A Phase II Study of Lenalidomide, Ixazomib, Dexamethasone, and Daratumumab in Transplant-Ineligible Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study of Lenalidomide/Ixazomib/Dexamethasone/Daratumumab in Transplant-Ineligible Patients With Newly Diagnosed MM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Celgene Corporation (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-41
Record Dates: First submitted 2019-06-20; First posted 2019-07-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Myeloma, Multiple
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; ixazomib; daratumumab; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenalidomide (Experimental): 12 cycles of lenalidomide, ixazomib, daratumumab, and dexamethasone followed by lenalidomide until disease progression or unacceptable toxicity or a maximum of 2 years of maintenance therapy.
  Interventions: Drug: Lenalidomide; Drug: Ixazomib; Drug: Daratumumab Injection; Drug: Dexamethasone
- Lenalidomide, Ixazomib, Daratumumab, and Dexamethasone (Experimental): 12 cycles of lenalidomide, ixazomib, dexamethasone, and daratumumab followed by lenalidomide, ixazomib, and daratumumab until disease progression or unacceptable toxicity or a maximum of 2 year maintenance therapy.
  Interventions: Drug: Lenalidomide; Drug: Ixazomib; Drug: Daratumumab Injection; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Induction and Maintenance
  Other Names: Revlimid
Drug: Ixazomib — Induction and Only Maintenance Arm B
  Other Names: Ninlaro
Drug: Daratumumab Injection — Induction and Only Maintenance Arm B
  Other Names: Darzalex
Drug: Dexamethasone — Induction and Only Maintenance Arm B
  Other Names: Ozurdex

SUMMARY:
A randomized Phase II clinical trial will be conducted to assess the impact on progression free survival (PFS) with the addition of ixazomib and daratumumab to lenalidomide as a maintenance treatment following induction with lenalidomide, ixazomib, dexamethasone, and daratumumab.

Patients will be randomized to either:

Arm A: 12 cycles of lenalidomide, ixazomib, daratumumab, and dexamethasone followed by lenalidomide until disease progression or unacceptable toxicity or a maximum of 2 years of maintenance therapy.

Arm B: 12 cycles of lenalidomide, ixazomib, daratumumab and dexamethasone, followed by lenalidomide, ixazomib, and daratumumab until disease progression or unacceptable toxicity or a maximum of 2 years maintenance therapy.

DETAILED DESCRIPTION:
Induction Phase: 28-day treatment cycle. Treatment continues until disease progression or for a maximum of 12 cycles as follows:

Cycles 1-2:

* Lenalidomide - 15 mg PO QD on Days 1-21
* Ixazomib - 4 mg PO on Days 1, 8, 15
* Daratumumab Subcutaneous - 15mL/1800mg on Days 1, 8, 15, 22
* Dexamethasone - 20 mg PO on Days 1, 2, 8, 9, 15, 16, 22, 23; For participants ≥75, dexamethasone administered on days 1, 8, 15, 22

Cycles 3-6:

* Lenalidomide - 15 mg PO QD on Days 1-21
* Ixazomib - 4 mg PO on Days 1, 8, 15
* Daratumumab Subcutaneous - 15mL/1800mg on Days 1, 15
* Dexamethasone - 20 mg PO on Days 1, 2, 8, 9, 15, 16; For participants ≥75, dexamethasone administered on days 1, 8, 15

Cycles 7-12:

* Lenalidomide - 15 mg PO QD on Days 1-21
* Ixazomib - 4 mg PO on Days 1, 8, 15
* Daratumumab Subcutaneous - 15mL/1800mg on Day 1
* Dexamethasone - 20 mg PO on Days 1, 2, 8, 9, 15, 16; For participants ≥75, dexamethasone administered on days 1, 8, 15

Maintenance Phase: 28-day treatment cycle. Treatment continues until progression or a maximum of 2 years of maintenance treatment:

Arm A

• Lenalidomide - 10 mg PO QD on Days 1-21

Arm B

* Lenalidomide - 10 mg PO QD on Days 1-21
* Ixazomib - 3 mg (or last tolerated dose from the induction phase) PO on Days 1, 8, and 15
* Daratumumab Subcutaneous - 15mL/1800mg on Day 1
* Dexamethasone - 20mg PO on Day 1; Unless patient is ≥75 then 10mg po day 1

In the maintenance phase, dexamethasone, 20 mg PO orally or IV will be administered to patients as a pre-infusion medication prior to daratumumab dosing. When dexamethasone is reduced to 20 mg/week and is given as pre-infusion medication, patients may receive low-dose methylprednisolone (≤20 mg) orally (or equivalent in accordance with local standards) for the prevention of delayed IRRs as clinically indicated.

If the investigator wishes to continue the maintenance regimen at the end of the 2 years maintenance treatment, patients may continue current maintenance as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age.
2. Subject must have documented multiple myeloma:

   * Clonal bone marrow plasma cells ≥10% or biopsy-proven bony or extramedullary plasmacytoma
   * Following CRAB features and/or myeloma-defining events (MDEs):

     * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically:

       * Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL) OR
       * Renal insufficiency: creatinine clearance <40 mL per minute or serum creatinine >177 mol/L (>2 mg/dL) OR
       * Anemia: hemoglobin value of >2 g/dL below the lowest limit of normal, or a hemoglobin value <100 g/L OR
       * Bone lesions: one or more osteolytic lesion on skeletal radiography, CT, or PET/CT. If bone marrow has <10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement OR
     * OR any one or more of the following biomarkers of malignancy (MDEs):

       * Sixty percent (60%) or greater clonal plasma cells on bone marrow examination.
       * Serum involved/uninvolved free light chain ratio of 100 or greater, provided the absolute level of the involved light chain is at least 100 mg/L (A patient's involved free light chain, either kappa or lambda, is the one that is above the normal reference range; the uninvolved free light chain is the one that is typically in, or below, the normal range).
       * More than one focal lesion on MRI that is at least 5 mm or greater in size.
3. Measurable disease as defined by any of the following:

   * IgG myeloma: serum monoclonal paraprotein (M-protein) level ≥0.5 g/dL; or
   * IgA, IgM, or IgD multiple myeloma: serum M-protein level ≥0.5 g/dL; or
   * Urine M-protein level ≥200 mg/24 hours; or
   * Serum free light chain ≥100 mg/L and abnormal serum immunoglobulin kappa lambda free light chain ratio
4. Newly diagnosed and not considered candidate for high-dose chemotherapy with stem cell transplant due to:

   * Age ≥70 years, OR
   * In patients <70 years: presence of important comorbid condition(s) likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation (ASCT) and/or site investigator's discretion due to concern regarding acute and long-term toxicity.
5. Patient must have an ECOG performance status score of 0, 1, or 2.
6. Patient must have adequate pretreatment clinical laboratory values meeting the following criteria ≤14 days of registration date:

   * Hemoglobin ≥7.5 g/dL (prior red blood cell transfusion or recombinant human erythropoietin use is permitted).
   * Absolute neutrophil count (ANC) ≥1x109/L (granulocyte colony stimulating factor (GCSF use is permitted).
   * Platelet count ≥75x109/L for patients in whom <50% of bone marrow nucleated cells are plasma cells; otherwise, platelet count >50×109/L (transfusions are not permitted to achieve this minimum platelet count).
   * Aspartate aminotransferase (AST) ≤3xULN.
   * Alanine aminotransferase (ALT) ≤3xULN.
   * Total bilirubin ≤1.5xULN, except in patients with congenital bilirubinemia, such as Gilbert syndrome (direct bilirubin ≤2xULN).
   * Creatinine clearance (CrCl) ≥30 mL/min. (Creatinine clearance may be calculated using the Cockcroft-Gault formula
   * Corrected serum calcium ≤14 mg/dL (≤3.5 mmol/L); or free ionized calcium <6.5 mg/dL (<1.6 mmol/L).
7. Women of childbearing potential (WOCBP) must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to initial dosing. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy. A man who is sexually active with a WOCBP must agree to use a latex or synthetic condom, even if they had a successful vasectomy. All men must also not donate sperm during the study, for 4 weeks after the last dose of lenalidomide, and for 4 months after the last dose of daratumumab. A WOCBP must have 2 negative serum or urine pregnancy tests first within 10 to 14 days prior to the registration date.
8. All study patients must be registered into the mandatory Revlimid REMS program and be willing and able to comply with the requirements of the REMS program.
9. Females of reproductive potential must agree to adhere to the scheduled pregnancy testing as required in the Revlimid REMS program.
10. At the time of registration, confirmation of adequate contraceptive method(s) should be documented in the medical record.
11. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Patient has primary AL amyloidosis.
2. Prior history of Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
3. Prior or current systemic therapy or stem cell transplantation (SCT) for MM, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before initial dosing. 1 cycle or less of urgent systemic treatment may be allowed after discussion with the Study Chair.
4. Patients undergoing treatment for a malignancy within 5 years prior to study enrollment with the exception of non-invasive malignancies that in the opinion of the site investigator are considered cured or have minimal risk of recurrence within 5 years. Patient must not have active concomitant, invasive malignancy. Note: patients on chronic hormonal therapy for localized breast or prostate cancer with no evidence for the primary malignancies or prostate cancer undergoing active surveillance can be included.
5. Radiation therapy ≤14 days prior to C1D1.
6. Plasmapheresis ≤28 days prior to C1D1.
7. Exhibiting clinical signs of meningeal involvement of MM ≤28 days prior to screening.
8. Known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume [FEV] in 1 second <60% of predicted normal), persistent asthma, or a history of asthma ≤ 2 years prior to screening (intermittent asthma is allowed).

   Note: Patients with known or suspected COPD or asthma must have a FEV1 test within 28 days prior to screening.
9. Patient has history or evidence of unstable/uncontrolled medical or psychiatric disorder, condition or disease (e.g., active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results, or that in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion.
10. Clinically significant cardiac disease, including:

    * myocardial infarction ≤1 year prior to screening, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV).
    * uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 5.0 Grade ≥2) or clinically significant ECG abnormalities;
    * 12-lead ECG performed ≤28 days prior to screening showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
11. Known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies, or human proteins, or their excipients (refer to respective package inserts or Investigator's Brochure) or known sensitivity to mammalian-derived products.
12. History of plasma cell leukemia (by WHO criterion: ≥20% of cells in the peripheral blood with an absolute plasma cell count of more than 2×10^9/L) or POEMS syndrome (ie, polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
13. Patient is:

    * seropositive for human immunodeficiency virus (HIV)
    * seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
    * seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
14. A woman who is pregnant, or breast-feeding, or planning to become pregnant during the study period or a man who plans to father a child during the study period. See Section 12.8 for further details.
15. Major surgery ≤14 days prior to screening or has not fully recovered from surgery, or has surgery planned during the time the patient is expected to participate in the study.

    Note: Kyphoplasty or vertebroplasty is not considered major surgery.
16. Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device ≤28 days prior to initial dosing or is currently enrolled in an interventional investigational study.
17. Contraindications to required protocol prophylaxis for deep vein thrombosis and pulmonary embolism.
18. Peripheral neuropathy Grade 2 or severe ≤28 days prior to screening.
19. Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort ≤14 days prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Impact of Study Treatment on Progression Free Survival (PFS) | 5 Years
  Time interval between registration and progression or death.

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) | 5 Years
  Minimal residual disease (MRD) negativity in the blood and marrow will be determined using the IMWG criteria.
Toxicity Profile of Treatment Arm Based on Patient Response | 5 Years
  Evaluation of incidence and severity of adverse events by summaries of toxicity data/contingency tables.
Overall Response Rate (ORR) | 5 Years
  Proportion of patients with reduction in tumor burden of a predefined amount.
Overall Survival (OS) | 5 Years
  Time from registration to death due to any cause.
Quality of Life with the EQ 5D 5L Questionnaire | 5 Years
  Consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Quality of Life with the EORTC QLQ-MY20 Questionnaire | 5 Years
  The EORTC QLQ-MY20 module was developed as an addition to the QLQ-C30 for use specifically in MM. It has 4 domains (disease symptoms, side effects of treatment, body image, future perspectives). Scores range from 0 to 100; good HRQoL is indicated by high scores for future perspective and body image, and low scores for disease symptoms and side effects of treatment.
Quality of Life with the EORTC QLQ-C30 Questionnaire | 5 Years
  The EORTC QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status/QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Rate of Adherence to Lenalidomide and Ixazomib | 5 Years
  All patients who have begun treatment will be included in the estimate of adherence rate to lenalidomide and the estimate of the adherence rate to ixazomib.
Alliance Geriatric Assessment with IMWG Fragility Score | 5 Years
  To describe functional status, comorbidity, psychological state, social activity, social support, chemotherapy toxicity, and nutrition using the geriatric assessment tool.

OTHER OUTCOMES:
Changes in Body Composition After Induction Therapy | 5 Years
  Fat and lean mass will be measured using dual energy X-ray absorptiometry (DXA previously DEXA).
Circulating MM cells and circulating DNA through DNA sequencing | 5 Years
  Blood samples will be collected to study DNA of normal and any potential tumor cells in blood. Further assessment of the genes, the RNA, and the proteins that are found in MM cells as well as in normal, noncancerous cells will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Principal Investigator — Alliance Foundation Trials, LLC.; Andrew Yee, MD, Study Chair — Massachusetts General Hospital
Locations (7):
- United States (7):
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - SUNY Upstate Medical Center, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Gibbs Cancer Center & Research Institute/Spartanburg Regional Healthcare, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Kyle RA, Gertz MA, Witzig TE, Lust JA, Lacy MQ, Dispenzieri A, Fonseca R, Rajkumar SV, Offord JR, Larson DR, Plevak ME, Therneau TM, Greipp PR. Review of 1027 patients with newly diagnosed multiple myeloma. Mayo Clin Proc. 2003 Jan;78(1):21-33. doi: 10.4065/78.1.21. PMID 12528874
- [Background] Kumar SK, Dispenzieri A, Lacy MQ, Gertz MA, Buadi FK, Pandey S, Kapoor P, Dingli D, Hayman SR, Leung N, Lust J, McCurdy A, Russell SJ, Zeldenrust SR, Kyle RA, Rajkumar SV. Continued improvement in survival in multiple myeloma: changes in early mortality and outcomes in older patients. Leukemia. 2014 May;28(5):1122-8. doi: 10.1038/leu.2013.313. Epub 2013 Oct 25. PMID 24157580
- [Background] Facon T, Mary JY, Pegourie B, Attal M, Renaud M, Sadoun A, Voillat L, Dorvaux V, Hulin C, Lepeu G, Harousseau JL, Eschard JP, Ferrant A, Blanc M, Maloisel F, Orfeuvre H, Rossi JF, Azais I, Monconduit M, Collet P, Anglaret B, Yakoub-Agha I, Wetterwald M, Eghbali H, Vekemans MC, Maisonneuve H, Troncy J, Grosbois B, Doyen C, Thyss A, Jaubert J, Casassus P, Thielemans B, Bataille R; Intergroupe Francophone du Myelome (IFM) group. Dexamethasone-based regimens versus melphalan-prednisone for elderly multiple myeloma patients ineligible for high-dose therapy. Blood. 2006 Feb 15;107(4):1292-8. doi: 10.1182/blood-2005-04-1588. Epub 2005 Sep 20. PMID 16174762
- [Background] Benboubker L, Dimopoulos MA, Dispenzieri A, Catalano J, Belch AR, Cavo M, Pinto A, Weisel K, Ludwig H, Bahlis N, Banos A, Tiab M, Delforge M, Cavenagh J, Geraldes C, Lee JJ, Chen C, Oriol A, de la Rubia J, Qiu L, White DJ, Binder D, Anderson K, Fermand JP, Moreau P, Attal M, Knight R, Chen G, Van Oostendorp J, Jacques C, Ervin-Haynes A, Avet-Loiseau H, Hulin C, Facon T; FIRST Trial Team. Lenalidomide and dexamethasone in transplant-ineligible patients with myeloma. N Engl J Med. 2014 Sep 4;371(10):906-17. doi: 10.1056/NEJMoa1402551. PMID 25184863
- [Background] Richardson PG, Weller E, Lonial S, Jakubowiak AJ, Jagannath S, Raje NS, Avigan DE, Xie W, Ghobrial IM, Schlossman RL, Mazumder A, Munshi NC, Vesole DH, Joyce R, Kaufman JL, Doss D, Warren DL, Lunde LE, Kaster S, Delaney C, Hideshima T, Mitsiades CS, Knight R, Esseltine DL, Anderson KC. Lenalidomide, bortezomib, and dexamethasone combination therapy in patients with newly diagnosed multiple myeloma. Blood. 2010 Aug 5;116(5):679-86. doi: 10.1182/blood-2010-02-268862. Epub 2010 Apr 12. PMID 20385792
- [Background] Kumar SK, Berdeja JG, Niesvizky R, Lonial S, Laubach JP, Hamadani M, Stewart AK, Hari P, Roy V, Vescio R, Kaufman JL, Berg D, Liao E, Di Bacco A, Estevam J, Gupta N, Hui AM, Rajkumar V, Richardson PG. Safety and tolerability of ixazomib, an oral proteasome inhibitor, in combination with lenalidomide and dexamethasone in patients with previously untreated multiple myeloma: an open-label phase 1/2 study. Lancet Oncol. 2014 Dec;15(13):1503-1512. doi: 10.1016/S1470-2045(14)71125-8. Epub 2014 Nov 14. PMID 25456369
- [Background] Lokhorst HM, Plesner T, Laubach JP, Nahi H, Gimsing P, Hansson M, Minnema MC, Lassen U, Krejcik J, Palumbo A, van de Donk NW, Ahmadi T, Khan I, Uhlar CM, Wang J, Sasser AK, Losic N, Lisby S, Basse L, Brun N, Richardson PG. Targeting CD38 with Daratumumab Monotherapy in Multiple Myeloma. N Engl J Med. 2015 Sep 24;373(13):1207-19. doi: 10.1056/NEJMoa1506348. Epub 2015 Aug 26. PMID 26308596
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Dredge K, Horsfall R, Robinson SP, Zhang LH, Lu L, Tang Y, Shirley MA, Muller G, Schafer P, Stirling D, Dalgleish AG, Bartlett JB. Orally administered lenalidomide (CC-5013) is anti-angiogenic in vivo and inhibits endothelial cell migration and Akt phosphorylation in vitro. Microvasc Res. 2005 Jan;69(1-2):56-63. doi: 10.1016/j.mvr.2005.01.002. PMID 15797261
- [Background] Corral LG, Haslett PA, Muller GW, Chen R, Wong LM, Ocampo CJ, Patterson RT, Stirling DI, Kaplan G. Differential cytokine modulation and T cell activation by two distinct classes of thalidomide analogues that are potent inhibitors of TNF-alpha. J Immunol. 1999 Jul 1;163(1):380-6. PMID 10384139
- [Background] Schafer PH, Gandhi AK, Loveland MA, Chen RS, Man HW, Schnetkamp PP, Wolbring G, Govinda S, Corral LG, Payvandi F, Muller GW, Stirling DI. Enhancement of cytokine production and AP-1 transcriptional activity in T cells by thalidomide-related immunomodulatory drugs. J Pharmacol Exp Ther. 2003 Jun;305(3):1222-32. doi: 10.1124/jpet.102.048496. Epub 2003 Mar 20. PMID 12649301
- [Background] Davies FE, Raje N, Hideshima T, Lentzsch S, Young G, Tai YT, Lin B, Podar K, Gupta D, Chauhan D, Treon SP, Richardson PG, Schlossman RL, Morgan GJ, Muller GW, Stirling DI, Anderson KC. Thalidomide and immunomodulatory derivatives augment natural killer cell cytotoxicity in multiple myeloma. Blood. 2001 Jul 1;98(1):210-6. doi: 10.1182/blood.v98.1.210. PMID 11418482
- [Background] Hideshima T, Chauhan D, Shima Y, Raje N, Davies FE, Tai YT, Treon SP, Lin B, Schlossman RL, Richardson P, Muller G, Stirling DI, Anderson KC. Thalidomide and its analogs overcome drug resistance of human multiple myeloma cells to conventional therapy. Blood. 2000 Nov 1;96(9):2943-50. PMID 11049970
- [Background] Richardson PG, Schlossman RL, Weller E, Hideshima T, Mitsiades C, Davies F, LeBlanc R, Catley LP, Doss D, Kelly K, McKenney M, Mechlowicz J, Freeman A, Deocampo R, Rich R, Ryoo JJ, Chauhan D, Balinski K, Zeldis J, Anderson KC. Immunomodulatory drug CC-5013 overcomes drug resistance and is well tolerated in patients with relapsed multiple myeloma. Blood. 2002 Nov 1;100(9):3063-7. doi: 10.1182/blood-2002-03-0996. PMID 12384400
- [Background] Richardson PG, Blood E, Mitsiades CS, Jagannath S, Zeldenrust SR, Alsina M, Schlossman RL, Rajkumar SV, Desikan KR, Hideshima T, Munshi NC, Kelly-Colson K, Doss D, McKenney ML, Gorelik S, Warren D, Freeman A, Rich R, Wu A, Olesnyckyj M, Wride K, Dalton WS, Zeldis J, Knight R, Weller E, Anderson KC. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006 Nov 15;108(10):3458-64. doi: 10.1182/blood-2006-04-015909. Epub 2006 Jul 13. PMID 16840727
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Background] O'Donnell EK, Laubach JP, Yee AJ, Chen T, Huff CA, Basile FG, Wade PM, Paba-Prada CE, Ghobrial IM, Schlossman RL, Burke JN, Harrington CC, Lively KJ, Lyons HF, Munshi NC, Anderson KC, Trippa L, Richardson PG, Raje NS. A phase 2 study of modified lenalidomide, bortezomib and dexamethasone in transplant-ineligible multiple myeloma. Br J Haematol. 2018 Jul;182(2):222-230. doi: 10.1111/bjh.15261. Epub 2018 May 8. PMID 29740809
- [Background] Hurria A, Cirrincione CT, Muss HB, Kornblith AB, Barry W, Artz AS, Schmieder L, Ansari R, Tew WP, Weckstein D, Kirshner J, Togawa K, Hansen K, Katheria V, Stone R, Galinsky I, Postiglione J, Cohen HJ. Implementing a geriatric assessment in cooperative group clinical cancer trials: CALGB 360401. J Clin Oncol. 2011 Apr 1;29(10):1290-6. doi: 10.1200/JCO.2010.30.6985. Epub 2011 Feb 28. PMID 21357782
- [Background] Hurria A, Togawa K, Mohile SG, Owusu C, Klepin HD, Gross CP, Lichtman SM, Gajra A, Bhatia S, Katheria V, Klapper S, Hansen K, Ramani R, Lachs M, Wong FL, Tew WP. Predicting chemotherapy toxicity in older adults with cancer: a prospective multicenter study. J Clin Oncol. 2011 Sep 1;29(25):3457-65. doi: 10.1200/JCO.2011.34.7625. Epub 2011 Aug 1. PMID 21810685
- [Background] Hurria A, Jones L, Muss HB. Cancer Treatment as an Accelerated Aging Process: Assessment, Biomarkers, and Interventions. Am Soc Clin Oncol Educ Book. 2016;35:e516-22. doi: 10.1200/EDBK_156160. PMID 27249761
- [Background] Hurria A, Gupta S, Zauderer M, Zuckerman EL, Cohen HJ, Muss H, Rodin M, Panageas KS, Holland JC, Saltz L, Kris MG, Noy A, Gomez J, Jakubowski A, Hudis C, Kornblith AB. Developing a cancer-specific geriatric assessment: a feasibility study. Cancer. 2005 Nov 1;104(9):1998-2005. doi: 10.1002/cncr.21422. PMID 16206252
- [Background] Manasanch EE, Shah JJ, Lee HC, Weber DM, Thomas SK, Amini B, Feng L, Berkova Z, Hildebrandt M, Orlowski RZ. Bortezomib, lenalidomide, and dexamethasone with panobinostat for front-line treatment of patients with multiple myeloma who are eligible for transplantation: a phase 1 trial. Lancet Haematol. 2018 Dec;5(12):e628-e640. doi: 10.1016/S2352-3026(18)30174-1. PMID 30501870